CLINICAL TRIAL: NCT06136117
Title: Mpox, Biology, Outcome, Transmission and Epidemiology - Prospective Follow-up of High-risk Contacts
Brief Title: Monkeypox, Biology, Outcome, Transmission and Epidemiology -Prospective Follow-up of High-risk Contacts
Acronym: MBOTE-CONTACT
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Leidos Biomedical Research, Inc. (Industry); Alliance for International Medical Action (Other); University of California, Los Angeles (Other); Institut de Recherche pour le Developpement (Other Government); University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: 1657/22
Record Dates: First submitted 2023-05-04; First posted 2023-11-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Mpox
Keywords: Monkeypox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
With the MBOTE-CONTACT study, a detailed follow-up study of high-risk contacts of mpox patients will be done. The MBOTE-CONTACT study will be nested in the NIH-Funded PALM-007 clinical trial (NCT05559099) and the MBOTE project on mpox transmission. The study will take place in Maniema Province, Democratic Republic of Congo (DRC). Participants will be recruited among high-risk contacts of mpox patients included in the PALM-007 trial. Consenting contacts will be either followed daily at the central study site or visited weekly by an outreach team in the community. They will be examined daily for signs and symptoms and asked to provide daily saliva and weekly blood samples for polymerase chain reaction (PCR) and/or serology. If participants develop mpox, they are offered treatment and enrollment in the PALM-007 trial.

ELIGIBILITY:
Inclusion Criteria:

* ▪ Be a high-risk contact of a laboratory-confirmed mpox case, with high-risk defined as having at least one the following types of exposure:
* living in the same household as an mpox patient
* having had sexual contact or intercourse with an mpox patient
* sleeping in the same room as an mpox patient
* sharing a meal with an mpox patient
* children: having played together

  * Last exposure to the mpox index case of less than 14 days ago
  * Patients of any age and gender (children aged < 10 years are excluded from venous blood sampling)
  * Patient or culturally acceptable representative is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Having previously been diagnosed with mpox in the last 3 months
* Inability or unwillingness to comply with the proposed follow-up schedule

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will take place in parallel to the PALM007 clinical trial, which evaluates the safety and efficacy of tecovirimat for the treatment of mpox. The study will recruit in Tunda, Maniema Province as well as in Kole, Sankuru province. These are the two sites where the PALM-007 has started. The study may expand to other potential PALM007 study sites, including Boende (Tshuappa Province), depending on the case burden and epidemiological context.Participants will be recruited among high-risk contacts of laboratory-confirmed mpox cases included in the ongoing PALM007 trial.Participants will be recruited according to two strategic tracks centered around 1) the study center and 2) the community.
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Study human-to-human transmission of Mpox virus (MPXV) by determining the secondary attack rate (SAR) among high-risk contacts of index patients. | 21 days
  Proportion of high-risk contacts with a positive MPXV PCR on any sample within 21 days after inclusion.

SECONDARY OUTCOMES:
To determine the rate of seroconversion amongst high-risk contacts of index patients. | 21 days
  The proportion of high-risk contacts with seroconversion for mpox antibodies on day 21 compared to baseline.
To estimate the extent of asymptomatic shedding of MPXV. | 21 days
  PCR positivity in any sample (blood, saliva) among participants who do not have any symptoms at the moment of sampling, but develop symptoms later during follow-up.
To estimate the extent of presymptomatic shedding of MPXV. | 21 days
  PCR positivity in any sample (blood, saliva) among participants who do not have any symptoms at the moment of sampling, but develop symptoms later during follow-up.
To estimate the duration between start of viral shedding and the appearance of prodromal symptoms. | 21 days
  Time between PCR positivity in any sample and appearance of systemic symptoms: either adenopathy, fever or dysphagia.
To estimate the incubation period of MPXV. | 21 days
  Time from last exposure to first PCR positivity. Time from last exposure to appearance of any symptom. Time from last exposure to appearance of skin lesions.
To characterize the clinical presentation of symptomatic secondary cases. | 21 days
  Frequency, timing and type of signs and symptoms observed among participants with a positive PCR.
To evaluate risk factors for infection and/or symptomatic disease. | 21 days
  Number of contacts with positive PCR on any sample AND/OR symptomatic disease and one of the following factors:
  * Different types of contact with the index case
  * Exposure to the same animal reservoir as the index case
  * Being vaccinated against mpox
  * Sociodemographic factors
To evaluate the protective effect of previous small pox vaccinations against infection and/or symptomatic disease. | 21 days
  number of previous vaccinate contacts positive PCR on any sample AND/OR symptomatic disease.
To estimate the duration between start of viral shedding and the appearance of skin symptoms. | 21 days
  Time between PCR positivity in any sample and appearance of skin lesions.

OTHER OUTCOMES:
To evaluate pre- or asymptomatic infectiousness. | 21 days
  Number of PCR-positive samples from which MPXV can be cultured in cell culture.
To evaluate characteristics of the index cases that influence the risk of secondary infection. | 21 days
  Association between PCR positivity on any sample AND/OR symptomatic disease in the contact and characteristics of the index cases (included in PALM 007) including:
  * disease severity of the index case
  * site of PCR positivity of the index case
  * viral load in samples obtained from the index case
To evaluate genomic differences in MPXV strains isolated from index and secondary cases | 21 days
  Whole genome sequencing of MPXV strains from index and secondary cases

CONTACTS AND LOCATIONS:
Overall Officials: Laurens Liesenborghs, Prof., Principal Investigator — Institute of Tropical Medicine
Locations (1):
- Tunda, Tunda, Maniema Province, Democratic Republic of the Congo